CLINICAL TRIAL: NCT05097222
Title: Impact of Photobiomodulation on Objective, Physiological Measures of Brain Function in Individuals With Post-Concussion Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr George Medvedev (Industry)
Collaborators: MediTech International Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Dr George Medvedev, Sponsor-Investigator, HealthTech Connex Inc.
Organization: HealthTech Connex Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BioFlex_PCS_001
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Post-Concussive Syndrome, Chronic; Post-Concussion Syndrome; Mild Traumatic Brain Injury
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Study participants will be blinded to the PBMT treatment regimen they will receive. Participants will wear opaque goggles to blind them from seeing any light emitted from the LED arrays.
  A trained laser technician will provide treatment to the study participants. The laser clinician will be unblinded to the participant's treatment allocation. Assessments will be performed by an independent blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active PBMT (Experimental): Participants will receive 50minutes of PBMT, three times a week, for 8 weeks.
  Interventions: Device: BioFlex Dualport System
- Sham PBMT (Sham Comparator): Participants will receive 50minutes of Sham PBMT, three times a week, for 8 weeks. The Sham device will appear to function like the treatment device without providing any power intensity (0% power). At 0% power, no light is emitted from the LEDs.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: BioFlex Dualport System — The device consists of a laptop computer preprogrammed with the Bioflex® Practitioner+ Software, the Bioflex® DUO 180+ array pad that has 180 bicolour Light Emitting Diodes (LED) that emit red and near infrared light, and two laser probes, the LD-R 100 that emits red light, and the LD-I 200 that emits near infrared light.
  Other Names: Photobiomodulation
  Arms: Active PBMT
Device: Sham device — Control
  Arms: Sham PBMT

SUMMARY:
Photobiomodulation therapy (PBMT) uses light to influence the mitochondria of cells. PBMT of the brain enhances the metabolic capacity of neurons and stimulates anti-inflammatory, anti-apoptotic, and antioxidant responses, as well as neurogenesis and synaptogenesis. Its therapeutic role in disorders such as dementia and Parkinson's disease, as well as to treat stroke, brain trauma, and depression has gained increasing interest.

BioFlex is a form of PBMT consisting of light-emitting diodes (LEDs) and laser diodes. BioFlex utilizes red and near infrared light which penetrates tissues up to a certain tissue depth and studies have shown stimulates tissue growth and repair at the cellular level. PBMT has been proven useful for the treatment of soft tissue pain. Several studies have shown benefit in using PBMT in the treatment of certain neurological conditions, including chronic, mild traumatic brain injury (mTBI).

The purpose of this exploratory investigation, therefore, is to examine efficacy of BioFlex laser therapy on measures of brain function in patients suffering from PCS after mild-moderate, closed-head, traumatic brain injury cases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 19 years of age or older
2. Diagnosis of persistent post-concussional syndrome after ≥3 months of traumatic brain injury, based on the ICD-10 criteria. This diagnosis should be given to the patient from a clinical practitioner. ICD-10 clinical criteria require a history of TBI and the presence of three or more of the following eight symptoms: 1) headache, 2) dizziness, 3) fatigue, 4) irritability, 5) insomnia, 6) concentration or 7) memory difficulty, and 8) intolerance of stress, emotion, or alcohol.
3. Current pharmacologic management can remain stable throughout the protocol.
4. Fluent in English
5. Able to understand the informed consent form, study procedures and willing to participate in study.

Exclusion Criteria:

1. Malignant skin carcinoma within the treatment area (neck and cranium)
2. Intake of photosensitizing medication.
3. Prior history of PBMT therapy
4. Current diagnosis of severe anxiety (or score of ≥15 on the GAD-7), severe depression (or score of ≥20 on the PHQ-9), schizophrenia or bipolar disorder
5. History of other major neurological disorder (brain cancer, dementia, multiple sclerosis, stroke)
6. Diagnosed epilepsy or history of seizures not effectively controlled by medications
7. Exposed to an investigational drug or device 30 days prior to starting the study, or concurrent use of an investigational drug or device while enrolled in the study
8. Pregnant, suspected to be pregnant or planning to become pregnant during the study
9. Contraindicated for the NeuroCatch® Platform 2, including:

9.1. Requires the use of hearing aids or a cochlear implant 9.2. Diagnosed with tinnitus that is currently active 9.3. Has temporary damage to hearing (e.g. punctured ear drum) 9.4. Unable to detect a 740Hz tone played at 85dB in both ears. 9.5. Implanted pacemaker or implanted electrical stimulators 9.6. Metal or plastic implants in the skull, excluding dental/facial implants 9.7. Unhealthy scalp (apparent open wounds and/or bruised or weakened skin) 9.8. Previous exposure to the NeuroCatch® Platform 2 audio sequences in the last 3 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Response size of selected ERPs (N100, P300, N400) acquired using the NeuroCatch Platform 2 | Visit 1/Baseline to Visit 3/End of Treatment (8 weeks)
  Event-related potentials (ERPs)
Response timing of selected ERPs (N100, P300, N400) acquired using the NeuroCatch Platform 2 | Visit 1/Baseline to Visit 3/End of Treatment (8 weeks)
  Event-related potentials (ERPs)

SECONDARY OUTCOMES:
Number of adverse events | Visit 1/Baseline to Visit 3/End of Treatment (8 weeks)
  Frequency and severity of adverse events
Number of adverse device effects | Visit 1/Baseline to Visit 3/End of Treatment (8 weeks)
  Frequency and severity of adverse device effects
Pain Catastrophizing Scale Score | Visit 1/Baseline to Visit 3/End of Treatment (8 weeks)
  Mean, standard deviation, and assessment of variance. It is a 13-item scale, with a total range of 0 to 52. Higher scores are associated with higher amounts of pain catastrophizing.
Rivermead Post-Concussion Symptoms Questionnaire Score | Visit 1/Baseline to Visit 3/End of Treatment (8 weeks)
  Mean, standard deviation, and assessment of variance. Scored on a scale of 0-64 where higher scores reflect greater severity of post concussive symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Center for Neurology Studies, Surrey, British Columbia
  - Meditech Rehabilitation Centre, Etobicoke, Ontario